CLINICAL TRIAL: NCT06524336
Title: Host Immune Dynamics Following Seasonal Malaria Chemoprevention in African Children
Status: Active, not recruiting | Type: Observational
Sponsor: Malaria Consortium (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: MCUGSMC24001
Record Dates: First submitted 2024-07-11; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Malaria,Falciparum
Keywords: malaria; blood stage immunity; anti-disease immunity; SMC
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — filter paper, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to identify immune features linked to protection against malaria, examining variations by age and sex, and measuring changes in immune responses over time following seasonal malaria chemoprevention (SMC). The primary objectives are:

1. Thorough examination of antibody immune responses in individuals before and after one or more SMC rounds.
2. Thorough examination of both innate and adaptive cellular immune responses in people residing in areas with regular SMC use.

Participants will include children aged 3 to 59 months who have received at least two or three SMC rounds, as well as children aged 5 to 15 years with no prior SMC exposure.

Upon identifying participants, study details will be provided, and written informed consent obtained. Demographic and clinical information will be collected using standard case record forms, including previous SMC uptake and routine malaria control interventions. Information on SMC use will be obtained from SMC cards/existing medical records, detailing the number of cycles received, adherence, and general health condition, including previous diseases and EPI vaccine uptake.

Data Collection:

* Face-to-face interviews by trained research assistants.
* Clinical assessments, including temperature, weight, and mid-upper arm circumference (MUAC).
* Sickle cell status testing at enrolment via samples analyzed at the Molecular Research Laboratory (MOLAB).
* Hemoglobin measurement using a HemoCue analyzer.

Malaria Diagnosis:

* Blood samples collected for malaria diagnosis using rapid diagnostic tests (RDTs) and microscopy.
* RDTs, such as Paracheck Pf, will be performed according to manufacturer instructions, with results available within 15 minutes.
* Participants testing positive for malaria will receive a full course of antimalarial treatment and counselling to visit the nearest health facility if symptoms worsen.

Thick Blood Smears:

* New glass slides labelled with participant ID will be used for thick blood smears.
* Blood smears will be dried and stored in a cool, dust-free environment before transportation to central laboratories.
* Slides will be stained with 2% Giemsa for 30 minutes and evaluated for parasitemia and gametocytes, with densities calculated accordingly.

The study will help understand the immune responses to malaria and the efficacy of SMC in different age groups.

DETAILED DESCRIPTION:
This will be a prospective cohort study with participant enrolment done in two districts in the Karamoja sub region.

The study population will consist of children aged 3 to 59 months - the target age group for SMC. A representative sample of children in the 5-15 years age group to characterize immune dynamics and responses in this age group as a comparator age group will be enrolled as well.

Inclusion criteria

* Children aged 3 to 59 months and 5-15 years in the selected districts
* Provision of Informed consent by parents/caregivers

Exclusion criteria

• Children known to be immunosuppressed due to malnutrition, HIV or other chronic diseases

When participants are identified, further details about the study will be provided and written informed consent will be obtained. Demographic and clinical information will then be collected using standard case record forms. Information will be collected on previous uptake of SMC and routine use of malaria control interventions. Information on previous SMC use will be obtained through a review of SMC cards/existing medical records. This information will include number of cycles/rounds received, adherence to SMC medication at each of these cycles and number of SMC rounds. Information will also be collected on general health condition of the child including previous diseases and EPI vaccine uptake (verified by immunization card). All participants will be interviewed face-to-face by trained research assistants and will be asked a series of questions. This will be followed by clinical assessment that include measurement of temperature, weight and mid-upper arm circumference (MUAC).

At enrolment, sickle cell status will be ascertained via testing of samples at the Molecular Research laboratory (MOLAB). Venipuncture blood samples will be collected at enrolment for sickle cell testing and hemoglobin measurement. Hemoglobin analysis will be carried out using a drop of blood (approximately 0.2mls) from the EDTA sample collected. The test will be conducted using a battery-operated portable HemoCue analyzer (HemoCue, Anglom, Sweden) which provides a result within one minute.

All enrolled participants will have blood samples collected for malaria diagnosis using rapid diagnostic tests (RDTs) and microscopy. Samples will also be collected for molecular analysis as needed.

Paracheck Pf, from Orchid Biomedical System, India or any other type of RDTs recommended by the Ministry of Health will be used. RDTs will be performed according to the directions provided for the specific tests, using the blood transfer device and reagent provided by the manufacturer. Tests will be performed by study personnel, and results will be available within 15 minutes. The results of the RDT will be provided to the participant or their parent/guardian verbally, and will be recorded on the appropriate case record form. Participants who test positive for malaria will be provided a full course of antimalarial treatment and will also be counselled to go to the nearest health facility immediately if their illness worsens.

New glass slides, frosted at one end, will be used to make the thick blood smears. Before making the smears, the lab technician will appropriately label the glass slides at the frosted end with the participant ID. Thick blood smears will be made by placing a drop of blood in the middle of the slide. An applicator stick will be used to spread the blood into a spot of approximately 1 cm in diameter. The blood smear will be dried on a slide tray in an ideally dust-free environment. For study sites away from the coordinating center, slides will be kept at the study health facilities protected from excessive heat and light for no longer than 1 week to avoid auto-fixation. The slides will be kept in a slide box and stored in the coolest place possible. The blood slides will then be transported to designated central laboratories. Thick blood smears will be stained with 2% Giemsa for 30 minutes and will be evaluated for the presence of parasitaemia (asexual forms only) and gametocytes. Parasite and gametocyte densities will be calculated from thick blood smears by counting the number of asexual parasites and gametocytes, respectively, per 200 leukocytes (or per 500, if the count is less than 10 parasites or gametocytes per 200 leukocytes), assuming a leukocyte count of 8,000/µl. A thick blood smear will be considered negative when the examination of 100 high power fields does not reveal asexual parasites or gametocytes. For quality control, all slides will be read by a second microscopist and a third reviewer will settle any discrepant readings.

Each time a thick blood smear is obtained blood will also be collected onto filter paper. Samples will be collected by venipuncture or by finger-prick sampling. Filter paper (Whatman no 1, Whatman 3MM; Whatman, Maidstone, UK) will be pre-cut into individual squares and stapled to a thick card which will serve as its cover. Blood spots will be collected onto the filter paper in volumes of approximately 25 µl per blood spot (4 blood spots per sample). Filter paper samples will be labelled with bar codes on the covering cardboard and will be allowed to dry at ambient temperature and relative humidity before closing the card over the filter paper (like closing a matchbook). Filter paper samples will be transported from the field in zip lock bags and placed into a stock card filter paper box for final storage at ambient temperature or at -20⁰C with a desiccant. Filter paper samples will be stored at our partner laboratory at IDRC in Kampala for future studies. Future molecular studies will be performed only for research purposes and will have no impact on the clinical management of study participants.

Molecular studies will include the extraction of DNA and/or RNA from filter paper, followed by characterization of parasite and host nucleic acid sequences using standard molecular procedures including PCR, DNA hybridization, restriction enzyme digestion, and/or nucleic acid sequencing. These will be performed at the CPHL laboratories where genomics capacity is already established.

Venipuncture blood samples will be collected aseptically by trained laboratory technologists. Approximately 6 mls of blood will be collected from children below 5 years and up to 10ml from children above 5 years in Heparin or EDTA tubes. This whole blood will be stored in either specific fixatives, including Paxgene reagent, used to assess cellular gene expression, and/or separated into plasma and peripheral blood mononuclear cells (PBMC) using a Ficoll gradient, following standard protocols. PBMC and plasma will be isolated from blood samples collected from enrolled participants at the central processing Laboratory at Moroto Hospital.

Whole blood collected in paxgene reagent will be stored at -80°C for whole blood transcriptomic studies. Plasma will be stored at -80°C for plasma-based immunologic studies, which will include measurement of levels of cytokines and other circulating inflammatory proteins (e.g., pro-inflammatory and anti-inflammatory cytokines), antibodies (e.g., malaria-specific antibodies), and/or other features related to the host immune response. PBMCs will be isolated by density gradient centrifugation (Ficoll-Histopaque; GE Life Sciences), counted, and cryopreserved in liquid nitrogen. PBMCs will be used to evaluate the innate and adaptive immune response e.g. malaria-specific T cell responses by flow cytometry, RNA sequencing, cytometry by time of flight (CyTOF), and/or other assays to assess the host immune response. Several of these assays utilizing PBMCs will be performed in our partner laboratories in Uganda. For all specimen types, two samples aliquots will be prepared, one for analysis in Uganda, and the other to be shipped to Stanford for additional immunology assays that are not available in Uganda.

De-identified plasma obtained from malaria-naïve, donors will be used as controls. For antibody functional assays (antibody-dependent cellular cytotoxicity or phagocytosis), large quantities of PBMCs for stimulation assays in immunology analyses will be obtained from blood bank donors at designated regional blood banks.

A comprehensive and longitudinal profiling of a broad array of host immune responses will be conducted to evaluate the impact of SMC on host immunity to malaria. To broadly profile the antibody response, a multiplex assessment of malaria-specific antibody responses will be performed using MagPix/Luminex, utilizing plasma collected from study participants in Uganda. Plasma antibody levels, subclass, and avidity will be measured, along with several additional Fc-dependent functional features of the antibody response, including complement fixation and antibody-dependent cellular cytotoxicity. The Luminex multiplex bead array assay to determine IgG levels, subclass, Fc receptor binding, and avidity against >18 pre-erythrocytic and blood-stage malarial antigens, including CSP, AMA-1, MSP1, MSP2, Rh5 and others will be performed at our collaborating partner laboratories in Kampala. In collaboration with partners at Stanford University (PI Jagannathan), the Luminex assay will be further optimized to study additional functional features of the antibody response. This includes complement fixation, antibody-dependent cellular cytotoxicity, and phagocytosis, which will be assessed as needed.

To comprehensively and longitudinally profile the innate and adaptive cellular immune responses in participants living in this area with sustained SMC, cellular phenotypes, function, and gene expression will be broadly measured from PBMCs collected from the same individuals over time. To study systems-level changes in cellular immune profiles in individuals, whole blood RNA sequencing will be performed using blood collected from Paxgene tubes, and plasma proteomics will be conducted using a nucleic-acid linked immune-sandwich assay. As these assays are not available in Uganda, they will be performed in the laboratory of collaborators at Stanford.

Multiparameter flow cytometry will be used to study innate and adaptive cellular phenotypes at the single-cell level. To study the functional response of individual immune cells, optimized stimulation assays with malaria antigens will be used. Phenotyping and functional assays will be conducted at a designated laboratory in Tororo or Kampala. In collaboration with partners at Stanford University (PI Jagannathan), additional assessments of the functional state of innate and adaptive immune cells will be performed, including epigenetics by time of flight (EpiTOF), single-cell RNA sequencing, and single-cell T and B cell receptor sequencing.

Plasma samples will also be stored for future In-depth analysis of the differential abundances of serum/plasma proteins which may help in identification of surrogate markers that and can provide valuable information regarding disease pathogenesis and host immune responses. This is important as there is currently a dearth of proteomic analysis in these settings.

All statistical analyses will be performed using STATA version 16 (College Station) or R version 4.2.0. Comparisons of cellular percentages between groups will be performed using the Wilcoxon rank sum and/or t test, and the Wilcoxon signed-rank and/or paired t test will be used to compare paired data. Associations between continuous variables will be assessed using Spearman's rank correlation. Two-sided p-values will be calculated for all test statistics and P < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 59 months and 5-15 years in the selected districts
* Provision of Informed consent by parents/caregivers

Exclusion Criteria:

* Children known to be immunosuppressed due to malnutrition, HIV or other chronic diseases

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will consist of children aged 3 to 59 months - the target age group for SMC. We will also enroll a representative sample of children in the 5-15 years age group to characterize immune dynamics and responses in this age group as a comparator age group.
  These children will be further categorized into different groups according to their previous exposure to SMC to include the following;
  * Group 1: Children with no prior intake of SMC (Katakwi district) - we will enroll a total of 40 children in this group in the two age categories (3 to 59 months and 5-15 years)
  * Group 2: Children who have received at least two rounds of SMC (Napak district) - we will enroll 130 children aged 3 to 59 months in this group
  * Group 3: Children who have received at least three rounds of SMC (Moroto district) - we will enroll 130 children aged 3 to 59 months in this group
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-10-28 (Estimated); Study Completion 2024-10-28 (Estimated)

PRIMARY OUTCOMES:
Antibody immune response | one year
  Number of study participants with protective antimalarial antibodies
Innate and adaptive immune responses | one year
  Number of study participants with cellular phenotypes and functions that are protective from malaria

SECONDARY OUTCOMES:
surrogate markers that predict risk of malaria | one year
  Number of individuals with surrogate markers that predict risk of malaria

CONTACTS AND LOCATIONS:
Locations (1):
- Moroto Hospital, Moroto, Karamoja, Uganda